CLINICAL TRIAL: NCT00289146
Title: Comparison of Immune Response Following Surgical Management of Renal Tumors
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kenneth Ogan, MD, Associate Professor, Emory University
Other Study IDs: 0021-2005
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Kidney Cancer
Keywords: kidney cancer, immunology
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Examine the effects of renal surgery on the immune system.

DETAILED DESCRIPTION:
Prospective study examining the effects of different surgical procedures on immune function. This may have bearing on overall cancer specific recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

* Kidney tumor patients scheduled for open or laparoscopic surgery

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open or laparoscopic surgeries for the treatment of kidney tumors.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ogan, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States